CLINICAL TRIAL: NCT04838470
Title: Looking for Prognostic Factors That Affect the Survival of Patients With Heart Failure
Brief Title: Prognosis Predictors for Heart Failure
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001285B0
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure; Rehabilitation; Morality; Hospitalization; Life Quality
Keywords: cardiac rehabilitation; multidisciplinary program; heart failure; mortality; renin-angiotensin-aldosterone system
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cardiac rehabilitation — multidisciplinary disease management program

SUMMARY:
This study is looking for the predictors of the survival or rehospitalization of patients with heart failure with reduced ejection fraction. Participants who are discharged from an acute heart failure hospitalization are enrolled.

DETAILED DESCRIPTION:
This study is looking for the predictors of the survival or rehospitalization of patients with heart failure with reduced ejection fraction. Participants who are discharged from an acute heart failure hospitalization are enrolled. The prognostic factors provide information about the treatment of this disease in the future. This study is a retrospective observational study. Investigators will collect data from May 2014 to July 2019 in the heart failure center of Kaohsiung Chang Gung Memorial Hospital. A follow-up is conducted at the Kaohsiung HF center until August 2020. Investigators want to know whether the risk factors such as atrial fibrillation, diabetes, nephropathy, and some biochemical indexes can be an index that predicts future survival or rehospitalization of these patients. Besides, investigators will also explore the cardiac rehabilitation can also effectively improve the survival rate of such patients.

ELIGIBILITY:
Inclusion Criteria:

* inpatient, age >= 20 years old, male or female
* patient with heart failure with a reduced ejection fraction and discharged alive from the hospital
* received heart failure disease management program

Exclusion Criteria:

* Estimated survival time < 6 months
* Long-term bedridden for more than 3 months
* Cannot tolerance exercise test due to muscular-skeletal disorder
* Cannot co-operate all functional studies
* Ventilator dependent
* Terminal heart status
* The family reject to participate in this project

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 792 patients were recruited between May 2014 and July 2019 and follow-up conducted at the Kaohsiung HF center until August 2020. All patients were introduced to a multidisciplinary HF disease management program (HFDMP).
Sampling Method: Non-Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | May, 2014 ~ August 2020
  Number of participants that had occurrence of the mortality which is defined as all-cause mortality

SECONDARY OUTCOMES:
first heart failure rehospitalization | May, 2014 ~ August 2020
  Number of Participants That Had Occurrence of the Endpoint, Which is Defined as First Heart Failure (HF) Hospitalization
Change From Baseline to Month 6 and Month 12 for the Kansas City Cardiomyopathy Questionnaire 12 (KCCQ 12) Clinical Summary Score | May , 2014 ~ August 2020
  Change from baseline to Month 6 and month 12 for the Kansas City Cardiomyopathy Questionnaire short form (KCCQ12) clinical summary score. KCCQ12 is a 12-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ12 clinical summary score is a composite assessment of physical limitations and total symptom scores.
  Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data sharing plan will be discussed with other investigators.